CLINICAL TRIAL: NCT07095998
Title: Evaluation of Nerve Excitability in Cisplatin-Induced Peripheral Neuropathy
Brief Title: Nerve Excitability in Cisplatin-Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ka-Wai Ho (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Ka-Wai Ho, Sponsor-Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-766
Record Dates: First submitted 2025-06-02; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy; Peripheral Neuropathy; Neurotoxicity Syndromes; Neuropathy
Keywords: Peripheral Neuropathy Due to Chemotherapy; Peripheral Neuropathy; Neurotoxicity Syndromes; Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neurotoxicity Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: Participants Without Cisplatin-Induced Peripheral Neuropathy (Experimental): 30 participants with no baseline neuropathy symptoms will be enrolled prior to starting cisplatin-based chemotherapy and will complete the following:
  * Baseline visit with neurological exams and conduction studies
  * Standard of care chemotherapy infusion (duration may vary depending on the chemotherapy regimen received)
  * Post-Infusion study visits via phone call (number of visits may vary depending on the chemotherapy regimen received)
  * In-clinic visit with neurological exams and conduction studies if participants develop cis-PN symptoms
    --If participants do not develop cis-PN symptoms, participants will be reevaluated 1 month post end of cisplatin treatment
  * 7-day end of treatment visit via phone call
  * 1-month post-treatment visit with neurological exams and conduction studies
  Interventions: Diagnostic Test: Threshold Tracking Nerve Conduction Studies
- Cohort B: Participants with Cisplatin-Induced Peripheral Neuropathy (Experimental): 30 participants with cis-PN symptoms will be enrolled and will complete the following:
  -One-time visit with neurological exams and conduction studies
  Interventions: Diagnostic Test: Threshold Tracking Nerve Conduction Studies

INTERVENTIONS:
Diagnostic Test: Threshold Tracking Nerve Conduction Studies — Measurement of nerve excitability parameters, including response to sub-threshold pre-pulses and other stimuli. The DS5 0 Isolated Bipolar Constant Current Stimulator is a non-invasive, non-therapeutic device that provides controlled electrical stimuli for detailed function assessment of the superficial radial, superficial peroneal, ulnar, and sural nerves.
  Other Names: TTNC; TTNCS

SUMMARY:
This study aims to evaluate nerve excitability in participants with cisplatin-induced peripheral neuropathy (cis-PN) using threshold tracking nerve conduction studies (TTNCS). By assessing changes in nerve excitability parameters, the study seeks to enhance understanding of the pathophysiology of cis-PN and identify early markers of neurotoxicity in participants undergoing cisplatin-based chemotherapy.

DETAILED DESCRIPTION:
This study aims to evaluate nerve excitability in participants with cisplatin-induced peripheral neuropathy (cis-PN) using threshold tracking nerve conduction studies (TTNCS). By assessing changes in nerve excitability parameters, the study seeks to enhance understanding of the pathophysiology of cis-PN and identify early markers of neurotoxicity in participants undergoing cisplatin-based chemotherapy.

Peripheral neuropathy is a sensory disorder where patients feel a burning, tingling, or pins-and-needles sensation in the hands and feet that can lead to oversensitivity or numbness.

The U.S. Food and Drug Administration (FDA) has not approved DS5 0 Isolated Bipolar Constant Current Stimulator as a diagnostic tool for Peripheral Neuropathy.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, questionnaires, and standard neurological exams called nerve conduction studies and Threshold tracking nerve conduction studies.

Participants will be placed into one of the following groups:

* Cohort A: Participants without previous treatment with cisplatin and are about to start treatment with Cisplatin.
* Cohort B: Participants with previous treatment with cisplatin in the past 3 months (and no longer being treated with cisplatin) and are currently experiencing cisplatin- induced peripheral neuropathy.

It is expected that about 60 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria Cohort A:

* Adults age ≥ 18 who will begin cisplatin-based chemotherapy either alone or in combination with other agents that are not known to cause neuropathy.
* Participants must have adequate hematologic parameters to allow chemotherapy.

Exclusion Criteria Cohort A:

* Pre-existing peripheral neuropathy;
* Family history of a genetic/familial neuropathy;
* Any contraindication for treatment with cisplatin as determined by their primary oncologist;
* Chemotherapy regimen combining cisplatin with another known chemotherapy agent that may cause peripheral neuropathy;
* Patients with cardiac or spinal stimulating devices;
* Women who are pregnant or breastfeeding;
* Adults with impaired consent capacity as patients must be able to fill out questionnaires regarding their neuropathy symptoms;
* Other medical conditions that in the opinion of the treating physician would make the protocol unreasonably hazardous for the patient;
* Patients not considered to be able to comply with the protocol.

Inclusion Criteria Cohort B:

* Adults age ≥ 18 with a diagnosis of cis-PN.
* The last dose of cisplatin must be ≥ 3 months prior to study enrollment. Patients who may have been previously enrolled in Cohort A of this study are eligible to participate in Cohort B if they continue to have cis-PN symptoms 3 months after completion of cisplatin therapy.

Exclusion Criteria Cohort B:

* Pre-existing peripheral neuropathy;
* Family history of a genetic/familiar neuropathy;
* History of cisplatin-based regimen combining cisplatin with another known chemotherapy agent that may cause peripheral neuropathy;
* Patients with cardiac or spinal stimulating devices;
* Women who are pregnant or breastfeeding;
* Adults with impaired consent capacity as patients must be able to fill out questionnaires regarding their neuropathy symptoms;
* Other medical conditions that in the opinion of the treating physician would make the protocol unreasonably hazardous for the patient;
* Patients not considered to be able to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of change in Nerve Excitability in comparison to baseline nerve excitability. | For Arm A, the time frame is at baseline and within 24 weeks of cisplatin initiation. For Arm B, the time frame is during the TTNCS procedure.
  Nerve excitability will be assessed via Threshold Tracking Nerve Conduction Study (TTNCS). Excitability parameters collected will include refractoriness, superexcitability, extent of threshold change in threshold electrotonus (hyperpolarizing 90-100ms). A composite excitability score is calculated to assess overall change in excitability parameters, all of which are weighted equally (Park, S.B., Lin, C.S.Y., Kiernan, M.C. Nerve Excitability Assessment in Chemotherapy-induced Neurotoxicity.J. Vis. Exp. (62), e3439, doi:10.3791/3439 (2012).

SECONDARY OUTCOMES:
Number of participants who develop neuropathy symptoms as assessed by CTCAE v. 5.0. | For Arm A, peripheral neuropathy symptoms will be assessed at baseline and the time of the development of Cis-PN symptoms over the course of 24 weeks. For Arm B, symptoms will be assessed immediately before the TTNCS procedure.
  The Wilcoxon signed rank test (two tailed) will be used to compared measurements at these time points.

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Wai Ho, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Tamar Berger, MD PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu